CLINICAL TRIAL: NCT02065648
Title: NATIVE Sequence for Non-Contrast MR Angiogram Compared With Conventional Contrast Enhanced 3D MRA on 3T Verio Magnet
Brief Title: Syngo NATIVE Contrast Enhanced 3D MRA on 3T Verio Magnet
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry)
Responsible Party: Principal Investigator, Rola Saouaf, MD, Director, Body and Cardiac MRI, Cedars-Sinai Medical Center
Other Study IDs: CSMC-2011-MR-02-01-NATIVE-Mos
Record Dates: First submitted 2014-01-17; First posted 2014-02-19 (Estimated); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Vascular Disease
Keywords: MRA; Syngo Native; Gadolinium; Non contrast
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Syngo NATIVE MRA: All consenting participants will receive an additional non-contrast Syngo NATIVE MRA sequence prior to contrast injection their standard of care MRA.

SUMMARY:
The purpose of the study is to compare non-contrast abdominal MR Angiogram (MRA) syngo NATIVE sequence performed on a 3T Verio Siemens magnet to a standard contrast-enhanced MRA performed as part of routine clinical care in patients with normal renal function to determine if the non-contrast NATIVE sequence is a viable alternative to contrast enhanced MRA in patients with renal insufficiency. There are no interventions--this is an observational study.

DETAILED DESCRIPTION:
If the NATIVE sequence proves to be a viable alternative to contrast enhanced MRA it will provide imaging physicians with the diagnostic tool to assess vascular disease in patients with renal insufficiency without placing them at risk for additional co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

Over age 18 Signed informed consent Referred for standard of care MRA

Exclusion Criteria:

No contra-indications for MRI/MRA ie implants which could interfere with magnets Renal insufficiency which would preclude use of contrast-enhanced contrast for a standard of care MRA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consenting patients referred for standard of care contrast-enhanced abdominal MR Angiography
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Effectiveness of non-contrast enhanced MRA sequence | 36 months
  Compare non-contrast enhanced MRA images with contrast-enhanced MRA images.

CONTACTS AND LOCATIONS:
Overall Officials: Rola Saouaf, MD, Principal Investigator — Cedars-Sinai Medical Center; Franklin G. Moser, MD, Study Director — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No